CLINICAL TRIAL: NCT06121700
Title: Radiotherapy, Chemotherapy and Anti-PD-1 Immunotherapy Followed by Surgical Resection in Patients With Limited Metastatic Gastric or Gastroesophageal Junction Adenocarcinoma: A Prospective, Single Arm, Phase II Trial
Brief Title: Radiotherapy + Chemoimmunotherapy Followed by Surgery in Patients With Limited Metastatic Gastric or GEJ Cancer
Acronym: Miracle-G
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Dazhi Xu, Professor, Chief Physician, Head of the First Department of Gastric Surgery, Fudan University Shanghai Cancer Center, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FDRT-2022-260-2977
Record Dates: First submitted 2023-10-19; First posted 2023-11-08 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Adenocarcinoma; Stomach Neoplasm; Gastroesophageal-junction Cancer; Oligometastatic Disease; Metastatic Cancer; Metastatic Gastric Cancer; Adenocarcinoma of the Stomach; Gastroesophageal Junction Adenocarcinoma; Metastatic Adenocarcinoma
Keywords: gastric cancer; GEJ Cancer; oligometastasis; limited metastatic; hypofractionated radiotherapy; immunotherapy; gastrectomy; metastasectomy
MeSH Terms: conditions — Adenocarcinoma; Stomach Neoplasms; Neoplasm Metastasis | interventions — spartalizumab; Trastuzumab; Drug Therapy; Metastasectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radiotherapy, Chemotherapy and anti-PD-1 Immunotherapy followed by Surgical Resection (Experimental): Participants will receive short course hypofractionated radiotherapy (HFRT) for the primary lesion, HFRT or stereotactic body radiotherapy (SBRT) for metastatic lesions, combined with systemic chemotherapy and anti-PD-1 immunotherapy. For patients with HER2-positive cancer (defined as IHC 3+ or 2+/ISH+), trastuzumab is used along with chemotherapy and anti-PD-1 antibody. Then, surgical resections of primary and metastatic lesions are performed as much as possible. For patients who need a widely invasive surgical approach or are inoperable, local ablative therapies such as radiofrequency ablation (RFA) and microwave ablation (MVA) can be alternatives. For patients undergoing surgical resections, postoperative treatment includes chemotherapy, which is determined by the researcher, and PD-1 antibody, which will be maintained until one year after surgery.
  Interventions: Radiation: Radiotherapy targeted to the primary lesion; Radiation: Radiotherapy targeted to the metastatic lesions; Biological: Anti-PD-1 monoclonal antibody; Biological: Trastuzumab; Drug: Chemotherapy; Procedure: R0 total/subtotal gastrectomy with D2 lymphadenectomy; Procedure: Metastasectomy; Procedure: Local ablative therapies

INTERVENTIONS:
Radiation: Radiotherapy targeted to the primary lesion — 5 to 7 fractions of short course hypofractionated radiotherapy (HFRT) targeted to the primary lesion.
Radiation: Radiotherapy targeted to the metastatic lesions — Hypofractionated radiotherapy (HFRT) or stereotactic body radiotherapy (SBRT) targeted to metastatic lesions. The target dose will be adjusted based on the lesion's site and diameter and organs at risk, with high-dose irradiation of 4-8 fractions. All metastatic lesions should be irradiated as much as possible, and partial lesion irradiation should be allowed when technically impractical.
Biological: Anti-PD-1 monoclonal antibody — The anti-PD-1 mAb is used on day 1 along with each cycle of chemotherapy. There are no restrictions on the choice of anti-PD-1 mAb. Patients can choose commonly used accessible monoclonal antibodies based on their personal preferences and financial status.
  The commonly used anti-PD-1 mAb usages are as follows: Nivolumab/Toripalimab 240mg solution intravenously once daily, Q2W. OR Nivolumab/Toripalimab 360mg solution intravenously once daily, Q3W; OR Pembrolizumab/Tislelizumab/Sintilimab/Camrelizumab, 200mg solution intravenously once daily, Q3W.
Biological: Trastuzumab — For patients with HER2-positive cancer (defined as IHC 3+ or 2+/ISH+), trastuzumab is used along with chemotherapy and anti-PD-1 antibody. The 3-weekly schedule of trastuzumab starts with a loading dose of trastuzumab of 8 mg/kg, followed by 6 mg/kg trastuzumab every 21 days.
  Other Names: Herceptin®
Drug: Chemotherapy — The investigator's choice of chemotherapy regimens included SOX, XELOX or FOLFOX. Their usages are as follows:
  SOX: S-1 twice a day, days 1-14, the dose of S-1 is accorded to body-surface area (BSA): patients with a BSA of less than 1.25 m2 receive 80 mg daily; those with a BSA of 1.25 m2 or more but less than 1.5 m2 receive 100 mg daily; and those with a BSA of 1.5 m2 or more receive 120 mg daily; and oxaliplatin 130 mg/m2, day 1, every 3 weeks; XELOX: Capecitabine 1000 mg/m2 twice a day, days 1-14 and oxaliplatin 130 mg/m2, day 1, every 3 weeks; FOLFOX: Leucovorin 400 mg/m2, day 1, fluorouracil 400 mg/m2, day 1 and 1200 mg/m2, days 1-2, and oxaliplatin 85 mg/m2, day 1, every 2 weeks.
Procedure: R0 total/subtotal gastrectomy with D2 lymphadenectomy — For patients with a good response to preoperative treatment, surgical resection of primary and metastatic lesions is recommended. For primary lesions, gastrectomy with standard D2 lymphadenectomy is commonly used. The type of gastrectomy performed depends on the location and extent of the primary lesion. For GEJ or upper-third tumors, a 3 cm esophageal margin is recommended, and a total gastrectomy or esophagogastrectomy is performed. For middle-third tumors, the gastric margin is recommended to be more than 5 cm, and total gastrectomy is performed. For lower-third tumors, a 2 cm duodenal margin is recommended, and subtotal or total gastrectomy is performed. Billroth I or Roux-en-Y gastrojejunostomy is performed for distal gastrectomy patients. Roux-en-Y esophagojejunostomy is performed for patients receiving total gastrectomy.
Procedure: Metastasectomy — For patients with a good response to preoperative treatment, surgical resection of primary and metastatic lesions is recommended. For metastatic lesions, the surgical procedure and resection range are determined by the surgeon.
Procedure: Local ablative therapies — Local ablative therapies such as radiofrequency ablation (RFA) and microwave ablation (MVA) achieve high rates of complete tumor eradication of small metastases, and can be seen as alternatives if a widely invasive surgical approach is required or patient is inoperable.

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy and safety of radiotherapy combined with chemotherapy and anti-PD-1 immunotherapy followed by surgery for the primary and metastatic lesions in patients with limited metastatic gastric or gastroesophageal junction adenocarcinoma. The main questions it aims to answer are: 1) If the multimodal treatment which includes anti-PD-1 immunotherapy and local therapies will improve the survival of this group of patients. 2) If the multimodal treatment which includes anti-PD-1 immunotherapy and local therapies can be performed safely in this group of patients.

Participants will receive short course hypofractionated radiotherapy (HFRT) for the primary lesion, HFRT or stereotactic body radiotherapy (SBRT) for metastatic lesions, combined with systemic chemotherapy and anti-PD-1 immunotherapy. For patients with HER2-positive cancer (defined as IHC 3+ or 2+/ISH+), trastuzumab is used along with chemotherapy and anti-PD-1 antibody. Then, surgical resections of primary and metastatic lesions are performed as much as possible. For patients who need a widely invasive surgical approach or are inoperable, local ablative therapies such as radiofrequency ablation (RFA) and microwave ablation (MVA) can be alternatives. For patients undergoing surgical resections, postoperative treatment includes chemotherapy, which is determined by the researcher, and PD-1 antibody, which will be maintained until one year after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Histopathologically confirmed adenocarcinoma of stomach (G) or gastroesophageal junction (GEJ) (excluding Siewert type I).
2. Limited metastatic status of disease.
3. At least one evaluable lesion in CT/MRI according to RESIST 1.1 is required.
4. The status of HER2 is clear.
5. pMMR/MSS confirmed by immunohistochemistry or gene test.
6. Male or female. Patient age ≥ 18 years and ≤ 75 years.
7. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) score of 0 or 1.
8. Physical state or organ function can tolerate the planned treatment of the study protocol, including systematic chemotherapy, immunotherapy with anti-PD-1 monoclonal antibody (mAb), primary lesion radiotherapy, metastatic lesion radiotherapy, and surgical resection of primary and/or metastatic lesions.
9. No previous surgery or antitumor therapies, including chemotherapy, radiotherapy, or immunotherapy, were administered.
10. Adequate hematological function: absolute neutrophil count (ANC) ≥ 1.5×109/L; platelet count ≥ 100×109/L; hemoglobin level ≥ 90 g/L.
11. Adequate hepatic function: total bilirubin ≤ 1.5×upper limit of normal (ULN); AST (SGOT) and ALT (SGPT) < 2.5 × ULN in the absence of liver metastases, or < 5 × ULN in case of liver metastases; ALP ≤ 2.5×ULN; ALB ≥ 30 g/L.
12. Adequate renal function: serum creatinine ≤ 1.5×ULN; creatinine clearance rate ≥ 60 ml/min.
13. Adequate coagulation function: INR/PT ≤ 1.5×ULN; APTT ≤ 1.5×ULN.
14. TSH is within the normal range; if TSH is out of the normal range, FT3 and FT4 should be investigated. If the test results of FT3/FT4 cannot be obtained, T3 and T4 can be accepted. 13. If the level of T3/T4 is normal, the patients can be selected.
15. Urine test: urine protein<2+; if the urine protein≥2+, the 24-hour urine protein quantification must be≤1g.
16. There is no serious concomitant disease, and the patient's life expectancy is more than 6 months.
17. Patients agree to sign written informed consent before recruitment.
18. Patients are willing and able to follow the protocol during the study, including receiving treatment and scheduled follow-up and examination.
19. Patients are willing to provide samples of blood and tissue.
20. Female patients should not be pregnant or breast feeding.
21. Female patients agree to take contraceptive measures during treatment and within 120 days after the last dose of anti-PD-1 mAb or 180 days after the last use of chemotherapy or radiotherapy.

Definition of the limited metastatic disease:

1. Retroperitoneal lymph node metastases (RPLM) only or at maximum one organ involved with or without RPLM.
2. There is no peritoneal seeding on diagnostic laparoscopy (P0).
3. The definition of RPLM includes but is not limited to para-aortal, intra-aorto-caval, parapancreatic or mesenteric lymph nodes. If the duodenum is invaded, retropancreatic nodes are not regarded as M1.
4. The definition of single organ metastasis in the study is as follows: a) Liver: maximum of 5 metastatic lesions that are potentially resectable and the metastases should be limited to one lobe and not involve important blood vessels or bile ducts. b) Lung: unilateral involvement, potentially resectable. c) Ovary: uni- or bilateral Krukenberg tumors in the absence of macroscopic peritoneal carcinomatosis. d) Adrenal gland: uni- or bilateral metastases. e) Extra-abdominal lymph node metastases, such as supraclavicular or cervical lymph node involvement. f) Bone: localized bone involvement (defined as being within one radiation field).
5. Other metastatic disease locations are considered, limited by the investigator and confirmed by the multidisciplinary team (MDT).

Exclusion Criteria:

1. Patients who have previously received surgery, chemotherapy, radiotherapy or immunotherapy for gastric cancer.
2. Patients have a history of cancer in the five years before enrollment except for squamous or basal cell carcinoma of the skin that was effectively treated and superficial bladder cancer, cervical carcinoma in situ and breast cancer in situ that was treated by operation.
3. Pregnant or lactating females or females planning to become pregnant or lactating. Women of childbearing age with a positive pregnancy test or without a pregnancy test in the baseline period. Menopausal women must have stopped menstruating for at least 12 months before being considered to have no chance of pregnancy.
4. Patients who had sexual activity (with the possibility of childbirth) and were unwilling to use contraception during the study period.
5. Patients with a history of allergies to any drugs that may be used in this study, including chemotherapy drugs.
6. History of allogeneic stem cell transplantation or organ transplantation.
7. Vaccinated with live vaccine within 28 days before recruitment.
8. Immunotherapy (interleukin, interferon, thymine) or other experimental treatment was given 28 days before enrollment.
9. History of anti-PD-1, PD-L1, PD-L2 or any other specific T-cell costimulation or checkpoint pathway targeted therapy.
10. History of using steroids (dose > 10 mg/d prednisone) or other systemic immunosuppressive therapy within 14 days before recruitment, except for patients treated with the following regimen: steroids used for hormone replacement (dose > 10 mg/d prednisone); local application of steroids with little systemic absorption; short-term (≤ 7 days) use of steroids to prevent allergy or vomiting.
11. Patients with weight loss of more than 20% within 2 months before recruitment.
12. Uncontrolled systemic diseases, including diabetes, hypertension, etc.
13. Uncontrollable pleural effusion, pericardial effusion, or ascites occurred within two weeks before recruitment.
14. Failure of important organs (heart, lung, liver, kidney, etc.).
15. Moderate or severe renal injury [creatinine clearance ≤ 50 ml/min (according to Cockcroft & Gault equation)], or SCR > ULN.
16. Dipyrimidine dehydrogenase (DPD) deficiency.
17. Patients with central nervous system (CNS) disorders or tumors, including brain metastases, peripheral nervous system disorders or psychiatric diseases.
18. Cerebrovascular accidents occurred within 6 months before recruitment.
19. Patients with peripheral neuropathy of NCI-CTCAE grade 1, except for those with disappearance of the deep tendon reflex.
20. Patients with a known history of uncontrolled or symptomatic angina, uncontrolled arrhythmias and hypertension, congestive heart failure, cardiac infarction or cardiac insufficiency within 6 months prior to study recruitment.
21. Pulmonary embolism occurred within 28 days before enrollment.
22. Patients who had the following history of pulmonary diseases: interstitial lung disease, noninfectious pneumonia, pulmonary fibrosis, or acute lung disease.
23. Patients with gastrointestinal bleeding or a high risk of bleeding within the first 2 weeks of enrollment.
24. Patients who experienced gastrointestinal perforation or fistula within 6 months prior to enrollment.
25. Upper gastrointestinal obstruction, dysfunction or malabsorption syndrome may affect the absorption of oral chemotherapy drugs.
26. Patients who cannot swallow or take medication orally.
27. Patients with a history of active autoimmune disease or refractory autoimmune disease.
28. Severe chronic or active infections requiring systemic antibiotics, antifungal or antiviral therapy, including tuberculosis and AIDS.
29. Known history of human immunodeficiency virus (HIV) infection.
30. Patients with untreated chronic hepatitis B or HBV-DNA exceeding 500 IU/ml or HCV-RNA positive.
31. Alcohol/drug abuse and medical, psychological or social conditions may interfere with patients' participation in the study or have an impact on the evaluation of the study results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | From the time of enrollment, assessed up to 5 years follow-up.
  The time from enrollment to death due to any reason.

SECONDARY OUTCOMES:
No evidence of disease (NED) rate | Assessed 1 year after treatment
  Rate of no evidence of disease for one year
Objective response rate (ORR) | From the time of enrollment, assessed up to 5 years follow-up.
  Proportion of patients with complete response (CR) or partial response (PR) to preoperative multimodal therapy. ORR will be evaluated using RESIST1.1 by CT/MRI of the chest, abdomen, and pelvis.
Progression-free survival (PFS) | From the time of enrollment, assessed up to 5 years follow-up.
  The time from enrollment to disease progression or death from any cause.
Toxicities | From the time of enrollment, assessed up to 28 days after the last dose of study therapy
  Number of participants with treatment-related adverse events (TrAEs) reported between the first dose and 28 days after the last dose of study therapy as assessed by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE), version 5.0.
Surgical morbidity | During or one month after surgery
  Surgery-related adverse events (SRAEs) refer to complications which happen during or one month after surgery. Severe complications after surgery will be documented and classified by Clavien-Dindo classification, such as abdominal or GI tract bleeding, anastomotic fistula, pancreatic fistula of grade B or above, and incision complications (infection, bleeding, rupture).
Surgical mortality | During or one month after surgery
  Death from any cause within 30 days of the date of surgery will be considered a surgical mortality death.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Al-Batran SE, Homann N, Pauligk C, Illerhaus G, Martens UM, Stoehlmacher J, Schmalenberg H, Luley KB, Prasnikar N, Egger M, Probst S, Messmann H, Moehler M, Fischbach W, Hartmann JT, Mayer F, Hoffkes HG, Koenigsmann M, Arnold D, Kraus TW, Grimm K, Berkhoff S, Post S, Jager E, Bechstein W, Ronellenfitsch U, Monig S, Hofheinz RD. Effect of Neoadjuvant Chemotherapy Followed by Surgical Resection on Survival in Patients With Limited Metastatic Gastric or Gastroesophageal Junction Cancer: The AIO-FLOT3 Trial. JAMA Oncol. 2017 Sep 1;3(9):1237-1244. doi: 10.1001/jamaoncol.2017.0515. PMID 28448662
- [Background] Al-Batran SE, Goetze TO, Mueller DW, Vogel A, Winkler M, Lorenzen S, Novotny A, Pauligk C, Homann N, Jungbluth T, Reissfelder C, Caca K, Retter S, Horndasch E, Gumpp J, Bolling C, Fuchs KH, Blau W, Padberg W, Pohl M, Wunsch A, Michl P, Mannes F, Schwarzbach M, Schmalenberg H, Hohaus M, Scholz C, Benckert C, Knorrenschild JR, Kanngiesser V, Zander T, Alakus H, Hofheinz RD, Roedel C, Shah MA, Sasako M, Lorenz D, Izbicki J, Bechstein WO, Lang H, Moenig SP. The RENAISSANCE (AIO-FLOT5) trial: effect of chemotherapy alone vs. chemotherapy followed by surgical resection on survival and quality of life in patients with limited-metastatic adenocarcinoma of the stomach or esophagogastric junction - a phase III trial of the German AIO/CAO-V/CAOGI. BMC Cancer. 2017 Dec 28;17(1):893. doi: 10.1186/s12885-017-3918-9. PMID 29282088
- [Background] Zhou ML, Xu RN, Tan C, Zhang Z, Wan JF. Advanced gastric cancer achieving major pathologic regression after chemoimmunotherapy combined with hypofractionated radiotherapy: A case report. World J Gastrointest Oncol. 2023 Jun 15;15(6):1096-1104. doi: 10.4251/wjgo.v15.i6.1096. PMID 37389115